CLINICAL TRIAL: NCT05167032
Title: A Clinical Trial of Cognitive Multisensory Rehabilitation for Sensory and Motor Recovery in Adults With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMR-2021-30498
Record Dates: First submitted 2021-12-20; First posted 2021-12-22 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Multisensory Rehabilitation (CMR) Group (Experimental): After the baseline testing, participants in the CMR group will receive 8 weeks of one-on-one, in-person therapy, 3 times a week, for 45 min. The CMR sessions will be recorded on video.
  The participants will undergo clinical assessments and MRI scans at 3 time points: at baseline; a post-intervention after the first 8 weeks of CMR and a clinical assessment (no MRI) at 3 months.
  Interventions: Behavioral: Cognitive Multisensory Rehabilitation (CMR)
- Adaptive Fitness Group (Active Comparator): After the baseline testing, participants in the adapted fitness group will start with a fitness assessment and then complete a fitness program under supervision for 8 weeks, 3x/week, for 45 min. Staff at the Courage Kenny Rehabilitation Institute will monitor training adherence through a log sheet.
  The participants will undergo clinical assessments and MRI scans at 3 times points: at baseline; a post-intervention after the first 8 weeks of adaptive fitness and a clinical assessment (no MRI) at 3 months.
  Interventions: Behavioral: Adaptive fitness

INTERVENTIONS:
Behavioral: Cognitive Multisensory Rehabilitation (CMR) — The goal of CMR is to restore proprioception (i.e., sense of joint position and movement), body awareness, and awareness of the paralyzed limbs and trunk in space, in order to improve sensory and motor function. For example, CMR tasks will have the participant solve exercises related to: (i) where the legs are situated in space; where the legs are in relation to the pelvis and the upper part of the body (ii) the dimensions and length of the legs, the dimension of the pelvis, and sensation of the pelvis as a central body reference. (iii) the relationship between the left and right side of the body, and the relationship between the pelvis and the feet. Further, improvements in touch and pressure sensation are obtained with (v) texture discrimination tasks, and (vi) discrimination of sponges with varying resistance. Given the importance of sensory feedback for movement, sensory improvements create the opportunity for motor recovery to occur.
  Arms: Cognitive Multisensory Rehabilitation (CMR) Group
Behavioral: Adaptive fitness — The Courage Kenny Rehabilitation Institute centers provide access to state-of- the-art adaptive gym equipment in their fitness center to promote fitness and recreation. Equipment includes treadmills, elliptical, NuSteps, SciFit upper body ergometers, Ski Erg and Rowing Machine, Upright and recumbent stationary bicycles, chest press, rear row, leg extension, leg curl, leg press, uppertone, free weights, and kettlebells. The equipment is spaced to allow for movement and is accessible for use from a wheelchair. They allow for transfers and caregiver assistance.
  Arms: Adaptive Fitness Group

SUMMARY:
To provide an effective treatment for recovery from paralysis and improved quality of life of veterans, military, and civilians with spinal cord injury/disorder (SCI/D). This is a mechanistic Phase I randomized pilot clinical trial in 16 adults with SCI/D. The investigators will compare the effects of Cognitive Multisensory Rehabilitation (CMR) vs. adaptive fitness on sensorimotor function. Objective 1: Determine if 8 weeks of CMR improves sensory and motor function in adults with SCI/D. Objective 2: Determine if 8 weeks of CMR restores brain activity and connectivity related to sensorimotor function in adults with SCI/D.

DETAILED DESCRIPTION:
About 296,000 Americans with a spinal cord injury/disorder (SCI/D) suffer from reduced or complete loss of sensory and motor function and 26% of adults with SCI receive care through the Veterans Affairs (VA). Motor and sensory impairments, including the loss of awareness of where limbs are in space, greatly compromise functional independence and quality of life. Damage to sensory and motor spinal pathways after SCI/D disrupts the bidirectional communication of sensory and motor information between the brain and the spinal cord, resulting in altered brain function in the sensorimotor cortex. Yet, an in-depth understanding of how exactly SCI/D impairs brain function, sensation and movement is largely unknown. Available treatments show mixed results for sensorimotor recovery, perhaps because it is unclear yet which specific brain areas to target. This highlights a need to develop brain mechanism-based treatments that restore brain function and improve sensation and movement after SCI/D. The investigators' brain imaging studies indicate that connections from two brain areas, the parietal operculum (parts OP1/OP4) and insula, are weaker in adults with SCI/D than in healthy adults. These connections are an essential part of the sensorimotor network. Thus, restoration of those network connections may lead to improved sensorimotor function after SCI/D. Previously, the investigators reported in adults 1-7 years post-stroke that OP1/OP4-insula connectivity restored alongside significantly improved sensorimotor function, by applying a physical therapy approach termed "Cognitive Multisensory Rehabilitation" (CMR). Based on these results, the investigators hypothesize that CMR restores brain connections related to sensorimotor function by strengthening OP1/OP4 and insula connections in adults with SCI/D. For this study, the investigators propose to test the hypothesis by carrying out the following objectives:

Objective 1: Determine if 8 weeks of CMR improves sensory and motor function in adults with SCI/D. The investigators will use quantitative measures used in clinical practice, and EMG testing to quantify changes in sensory and motor function. As secondary outcomes, the investigators will assess mood, life satisfaction, and community integration.

Hypothesis 1. CMR in comparison to adaptive fitness will improve sensorimotor function after SCI/D. Sensorimotor function will be associated with mood, life satisfaction, and community integration.

Objective 2: Determine if 8 weeks of CMR restores brain activity and connectivity related to sensorimotor function in adults with SCI/D. The investigators will assess changes in brain activation and connectivity in response to CMR vs adaptive fitness by resting-state and 4 task-based functional Magnetic Resonance Imaging (fMRI).

Hypothesis 2. CMR will restore OP1/OP4 and insula connectivity with other sensorimotor-related brain areas. These brain function changes will be associated with sensory and motor improvements.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete or complete SCI/D of ≥3 months
* Medically stable.

Exclusion Criteria:

* MRI contra-indications (stabilizing hardware is typically MRI safe)
* Uncontrolled seizure disorder
* Cognitive impairment and/or communicative disability (e.g., due to brain injury) that prevent individuals from following directions or from learning
* Ventilator dependency
* Other major medical complications
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Brain Motor Control Assessment (BMCA) | 3 Months
  The EMG testing will be done with the BMCA. The BMCA protocol involves elements of relaxation, reinforcement, and voluntary movements to gather quantitative multichannel surface EMG data. BMCA will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
  Assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
Change in ISNCSCI Neurologic exam (ASIA test) | 3 Months
  The ASIA test is a clinical test originally designed to describe the extent and severity of a patient's SCI/D. It consists of a pinprick sensory test (sharp versus dull with a safety pin); a touch sensory test (with a cotton ball) and a test of the strength of muscles. Each sensation test is scored from 0-54 right and left, and the muscle tests for upper and lower limbs are scored from 0-25 each. Higher scores indicate better function. The ASIA test will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
Change in Neuromuscular Recovery Scale (NRS) | 3 Months
  The NRS includes 11 items rated from 1-4 focused on the capacity of the trunk and lower extremity muscles to perform tasks such as sit, trunk extension, sit to stand, walking, and step retraining. Higher scores indicate better performance. The NRS provides a functional recovery measure that focuses on non-compensatory recovery. The NRS will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
Change in Spinal Cord Injury Functional Index/Assistive Technology (SCI-FI/AT) | 3 Months
  The SCI-FI/AT consists of 32 items each rated from 0-4, where higher scores indicate better function. It reliably measures function in the domains of basic mobility, self-care, fine motor function, and ambulation. The SCI-FI/AT will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
Change in International Spinal Cord Injury Pain Basic Set Version 2.0 (SCI Pain Test) which includes the numerical pain rating scale | 3 Months
  The SCI Pain Test consists of a numeric pain rating scale with scores ranging from 0-10 where lower scores indicate less pain, and an assessment of interference of pain with daily activity, mood, and sleep, with scores ranging from 0-10 where lower scores indicate less interference in daily life. The SCI Pain Test will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index | 3 Months
  The Pittsburgh Sleep Quality Index consists of 7 components with total scores ranging from 0-21, where lower scores indicate less difficulty in the assessed areas. The Pittsburgh Sleep Quality Index will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
Change in Spielberger State Trait Anxiety Inventory | 3 Months
  The Speilberger State Trait Anxiety Inventory consists of the trait anxiety scale which assesses general feeling and the state anxiety scale which assesses present feelings. Both scales are scored from 20-80, where lower scores indicate less anxiety.
  The Spielberger State Trait Anxiety Inventory will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
Change in Patient Health Questionnaire (PHQ-9) | 3 Months
  The PHQ-9 consists of 9 items scoring depression. Each item is scored from 0-3, with total scores ranging from 0-27, and higher scores indicate greater depressive symptoms. The PHQ-9 will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
Change in World Health Organization Quality of Life Instruments (WHOQOL-BREF) | 3 Months
  The WHOQOL-BREF is used to assess physical and psychological health, social relationships and environment. It consists of 4 domains assessed from 0-100, where higher scores indicate greater quality of life. The WHOQOL-BREF will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
Change in Revised Body Awareness Rating Questionnaire | 3 Months
  The Revised Body Awareness Rating Questionnaire is a 12-item scale assessing how tension in the body affects one's body awareness and function in daily life. Each item is scored from 0-3, with total scores ranging from 0-36. Lower scores indicate better body awareness. The Revised Body Awareness Rating Questionnaire will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
Change in Kinesthetic and Visual Imagery Questionnaire (KVIQ) | 3 Months
  The KVIQ assesses a 5-point ordinal scale the clarity of the image (visual) and a 5-point ordinal scale of the intensity of the sensations (kinesthetic) that the subjects are able to imagine from the first-person perspective imagery. Each item is scored 1-5 and summed for a global score, higher scores indicating better imagery. KVIQ will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
Change in Moorong Self-Efficacy Scale (MSES) | 3 Months
  The MSES consists of 16 items each scored from 1-7, with total global scores ranging from 16-112. The MSES assesses self-efficacy related to everyday life activities and is designed specifically for people with SCI/D. Higher scores indicate greater self-efficacy. The MSES will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
Change in Tampa Scale for Fear of Re-Injury | 3 Months
  The Tampa Scale consists of 17 items each scored from 1-4 with global scores ranging from 17-68. Lower scores indicate greater fear of re-injury. The Tampa Scale will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
Change in Patient-Specific Functional Scale | 3 Months
  For the Patient-Specific Functional Scale, the participant reports on 3 activities that are important to the participant that they are unable to do because of their pain. Participants rate them between 0 (unable to do the activity) and 10 (able to do the activity). The scale assesses perceived disability in adults with chronic conditions.
  The Patient-Specific Functional Scale will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.
The Craig Handicap Assessment and Reporting Technique-Short Form (CHART-SF) | 3 Months
  The CHART-SF assesses the degree by which a person with SCI/D remains with impairment or disability. It measures the type and level of assistance needed physically and cognitively; the level of physical activity; transportation needs; how time is spent; social interactions; and financial resources. Each of six domains is scored from 0-100, with total scores ranging from 0-600. Higher scores indicate less impairment. The CHART-SF will be assessed at baseline, 8 weeks after intervention, and during 3-month follow-up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Van de Winckel, PhD, MSPT, PT, Principal Investigator — University of Minnesota Medical School Department of Rehabilitation Medicine
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No